## <u>Official Title:</u> Amped-PD: Amplifying Physical Activity Through a Novel Digital Music Therapeutic in Parkinson Disease

**NCT#:** NCT05421624

**Date**: July 12, 2022

Statistical Analysis Plan (SAP)

## **Statistical Analysis Plan**

We will use parametric statistics to data with normal distribution verified using Shapiro-Wilk test and to data that meet the assumptions of homogeneity of variances using Levene's test. Otherwise, non-parametric statistics will be used.

To examine between-group differences for all primary outcomes (moderate intensity minutes, daily steps, stride time variability, and habit strength), we will run a one-way ANOVA or Kruskall-Wallis test to compare change scores at the 6-Week and 8-Week clinical assessments relative to baseline.

To examine within-group differences for all primary outcomes (moderate intensity minutes, daily steps, stride time variability, and habit strength), we will run a Repeated Measures ANOVA or Friedman's ANOVA on absolute values of all primary outcomes across their respective timepoints, with multiple post-hoc comparisons corrected using Bonferroni adjustments.

For all secondary outcomes, we will perform between-group analyses using non-parametric statistics to compare change scores at the 6-Week and 8-Week clinical assessments relative to baseline, using two-tailed tests with alpha set at 0.05.